CLINICAL TRIAL: NCT05386667
Title: Evaluation of the Effects of Medicaments Used After Free Gingival Graft on Postoperative Complications.
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, AYSAN LEKTEMUR ALPAN, Associate Profesor, Pamukkale University
Other Study IDs: 05.03.2019/05
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Pain, Postoperative; Healing Wound; Hemorrhage; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Hemorrhage; Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Control: Patients were not given anything after FGG.
  Interventions: Procedure: Free gingival graft harvesting
- Flurbiprofen: Oral spray containing 0.075 g flurbiprofen administered after FGG
  Interventions: Drug: Majezik %0.25 oral spray; Procedure: Free gingival graft harvesting
- Hypochlorous acid: Oral spray containing hypochlorous acid applied after FGG
  Interventions: Other: Crystalin oral spray; Procedure: Free gingival graft harvesting
- Hyaluronic acid: An oral spray containing the main component of the product is hyaluronic acid (sodium salt) with a high molecular weight of 30 mg / 100 g was given to patients after FGG
  Interventions: Other: Aftamed oral spray; Procedure: Free gingival graft harvesting

INTERVENTIONS:
Drug: Majezik %0.25 oral spray — Free gingival graft was taken from the palatal mucosa of the patients in order to increase the attached gingiva.
  After FGG, the patients were asked to apply this spray to the palatal mucosa 3 times a day.
  Other Names: Free gingival graft harvesting
  Groups: Flurbiprofen
Other: Aftamed oral spray — Free gingival graft was taken from the palatal mucosa of the patients in order to increase the attached gingiva.
  After FGG, the patients were asked to apply this spray to the palatal mucosa 3 times a day.
  Other Names: Free gingival graft harvesting
  Groups: Hyaluronic acid
Other: Crystalin oral spray — Free gingival graft was taken from the palatal mucosa of the patients in order to increase the attached gingiva.
  After FGG, the patients were asked to apply this spray to the palatal mucosa 3 times a day.
  Other Names: Free gingival graft harvesting
  Groups: Hypochlorous acid
Procedure: Free gingival graft harvesting — Free gingival graft was taken from the palatal mucosa of the patients in order to increase the attached gingiva.

SUMMARY:
In our study, three different medicaments were evaluated in terms of postoperative complications after free gingival grafting (FGG).

DETAILED DESCRIPTION:
In our study, three different medicaments were evaluated in terms of postoperative complications after free gingival grafting. The effectiveness of these 3 different commercially available agents containing flurbiprofen, hyaluronic acid, and hypochlorous acid, after use 2., 4.7. and on the 14th day, wound healing and pain perception was compared with the control group. primary observation was obtained by visual analog scale, wound healing index, bleeding of tissue, color match, and amount of painkiller used by the patient were also recorded

ELIGIBILITY:
Inclusion Criteria:- Patients with systematic conditions are classified as The American Society of Anesthesiologists Class I

-

Exclusion Criteria:

* Pregnancy, lactation, and taking contraceptive pills.
* Oversensitivity or anaphylactic reactions which contraindicate the intervention.
* Orofacial neurological symptoms.
* Infections at operation zone.
* Psychotropic medicine, sedative, or non-steroid anti-inflammatory drugs use which can alter the sense of pain.
* Pathological mental conditions (dementia, psychosis) and lack of cooperation.
* Smoking
* Excessive gag reflex
* Operations are carried out with conscious sedation.
* Patients who do not want to sign consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the study consists of all patients, who were planned to be applied free gingival graft for mucogingival surgery
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Landry's Wound Healing Index (WHI) | 21 days
  WHI was performed on the basis of postoperative healing characteristics categorized as tissue color, response to palpation, incision margins, and suppuration.

SECONDARY OUTCOMES:
Visual Analogue Scale | 21 days
  Recording the pain perception of the patients on a scale from 0 to 10. 0 - no pain 10 - worst pain
Color match | 21 days
  scoring the color match of the healed tissue area with the patient's remaining tissue
delayed bleeding | 21 days
  examining the patient whether there is postoperative bleeding, if there is a positive, if not, it should be recorded as negative.
burning sensation | 21 days
  Evaluation of the burning sensation felt in the healing area of the patient's palate from 0 to 10. 0-no burning sensation 10- excessive burning
complete epithelization | 21 days
  Examination of epithelialization with 3% oxygenated water. keeping records according to the foaming rate in the tissue

CONTACTS AND LOCATIONS:
Overall Officials: AYSAN LEKTEMUR ALPAN, PhD, Principal Investigator — Pamukkale Univesity
Locations (1):
- Pamukkale University Faculty of Dentistry Department of Periodontology, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We may share the obtained data personally, but the decision of this is not yet clear.

REFERENCES:
- [Background] Isler SC, Eraydin N, Akkale H, Ozdemir B. Oral flurbiprofen spray for mucosal graft harvesting at the palatal area: A randomized placebo-controlled study. J Periodontol. 2018 Oct;89(10):1174-1183. doi: 10.1002/JPER.17-0381. Epub 2018 Aug 29. PMID 30007054
- [Background] Hassan A, Ahmed E, Ghalwash D, Elarab AE. Clinical Comparison of MEBO and Hyaluronic Acid Gel in the Management of Pain after Free Gingival Graft Harvesting: A Randomized Clinical Trial. Int J Dent. 2021 Aug 14;2021:2548665. doi: 10.1155/2021/2548665. eCollection 2021. PMID 34426739
- [Background] Yildirim S, Ozener HO, Dogan B, Kuru B. Effect of topically applied hyaluronic acid on pain and palatal epithelial wound healing: An examiner-masked, randomized, controlled clinical trial. J Periodontol. 2018 Jan;89(1):36-45. doi: 10.1902/jop.2017.170105. PMID 28914592